CLINICAL TRIAL: NCT04848662
Title: A Phase I, Randomized, Open-label, Single-dose, 2-way Crossover Study to Compare the Pharmacokinetics of Budesonide Delivered by PT027 to Pulmicort Respules® in Children With Asthma Aged 4 to 8 Years (BLANC)
Brief Title: To Compare the Pharmacokinetics of Budesonide Delivered by BDA MDI to Budesonide Delivered by Pulmicort Respules in Children With Asthma Aged 4 to 8 Years.
Acronym: BLANC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bond Avillion 2 Development LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AV006
Record Dates: First submitted 2021-04-01; First posted 2021-04-19 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A/B - Treatment with BDA MDI (PT027) 160/180 μg followed by treatment with Pulmicort Respules 1mg (Experimental): Subjects randomized to receive a single dose of budesonide/albuterol by metered-dose inhaler, BDA MDI, (PT027) 160/180 μg at Visit 2, and a single dose of budesonide by nebulization (Pulmicort Respules) 1mg at Visit 3.
  Interventions: Drug: BDA MDI (PT027) 160/180 μg; Drug: Pulmicort Respules 0.5 MG/ML Inhalation Suspension
- B/A - Treatment with Pulmicort Respules 1 mg followed by treatment with BDA MDI (PT027) 160/180 μg (Experimental): Subjects randomized to receive a single dose of budesonide by nebulization (Pulmicort Respules) 1mg at Visit 2, and a single dose of budesonide/albuterol by metered-dose inhaler, BDA MDI, (PT027) 160/180 μg at Visit 3.
  Interventions: Drug: BDA MDI (PT027) 160/180 μg; Drug: Pulmicort Respules 0.5 MG/ML Inhalation Suspension

INTERVENTIONS:
Drug: BDA MDI (PT027) 160/180 μg — Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 80/90 μg per puff. Two puffs to administer 160/180 μg dose.
  Other Names: PT027
Drug: Pulmicort Respules 0.5 MG/ML Inhalation Suspension — Budesonide 0.5 mg/ml. Each 2 ml Respule contains 1 mg budesonide.

SUMMARY:
To compare the pharmacokinetics of budesonide delivered by BDA MDI to budesonide delivered by Pulmicort Respules in children with Asthma aged 4 to 8 years.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures. Children should provide assent to join the study, as applicable. The child's parent(s) or legally authorized representative (LAR) must sign the informed consent form (ICF). The LAR must be aged ≥18 years old.
2. Male or female aged between 4 and 8 years inclusive (not having reached his/her 9th birthday by the time of screening).
3. Weigh at least 14 kg or higher.
4. Clinician diagnosed asthma of at least 3 months.
5. Stable on treatment with albuterol PRN and/or ICS and/or leukotriene receptor antagonists (LTRAs) for 2 weeks prior to screening; children taking budesonide in any form at Visit 1 will be switched to another corticosteroid with a washout of budesonide of 3 to 7 days.
6. Demonstrate ability to correctly use the nebulizer and metered-dose inhaler (MDI) device without a spacer.
7. Willingness and ability of the child and parent(s)/LAR to comply with the demands of the study as described in the informed consent/assent.

Exclusion Criteria:

1. Inability to change from any budesonide therapy to another suitable corticosteroid.
2. History of life-threatening asthma defined as any asthma episode associated with loss of consciousness, intubation or admission to an intensive care unit.
3. Unstable asthma as judged by the Investigator (eg, any change in asthma therapy within 2 weeks prior to screening or use of more than 2 occasions of rescue medication (albuterol) per day within 1 week prior to screening (potential for rescreen).
4. Children receiving regular maintenance treatment with prohibited anti-inflammatory or long-acting bronchodilator asthma medication (inhaled, nebulized, oral, or systemic) within 1 month prior to screening.
5. More than 1 short course of oral/rectal/systemic corticosteroids within 6 months preceding screening (Visit 1), or any oral/rectal/systemic corticosteroids within 30 days prior to screening.
6. Evidence of active concomitant pulmonary disease other than asthma (children with stable allergic rhinitis will be permitted, as long as, there are no changes in the treatment and the medications do not interfere with the analytical assay methods).
7. Upper respiratory infection involving antibiotic treatment not resolved within 14 days prior to Visit 1.
8. Children with a known or suspected hypersensitivity to albuterol/salbutamol, budesonide or any of the excipients used in the IMPs.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Albers, MD, PhD, Study Director — Avillion LLP
Locations (2):
- United States (2):
  - IPS Research, Oklahoma City, Oklahoma
  - TTS Research, Boerne, Texas

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target population consisted of male or female children aged between 4 and 8 years who had clinician-diagnosed asthma of at least 3 months. Subjects were expected to be stable on treatment with albuterol as needed and/or inhaled corticosteroids and/or leukotriene receptor antagonists for 2 weeks prior to screening. The first subject enrolled on 06 May 2021 and the last subject completed the study on 08 July 2021. Subjects were enrolled at 2 US study centers.
Pre-assignment Details: The randomized treatment phase started after a screening period with a maximum duration of 14 days. Subjects who were taking budesonide in any form at Visit 1 were switched to another corticosteroid with a washout of budesonide of 3 to 7 days. In addition to the 12 subjects randomized, 1 subject was screened but did not participate (1 screen failure).
Groups:
- A/B - Treatment With BDA MDI (PT027) 160/180 μg Followed by Treatment With Pulmicort Respules 1mg: Subjects randomized to receive a single dose of budesonide/albuterol by metered-dose inhaler, BDA MDI, (PT027) 160/180 μg at Visit 2/Period 1, and a single dose of budesonide by nebulization (Pulmicort Respules) 1mg at Visit 3/Period 2.
  Visit 2/Period 1 (Day 1) - BDA MDI (PT027) 160/180 μg: Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 80/90 μg per puff. Two puffs to administer 160/180 μg dose.
  Visit 3/Period 2 (Day 8 +/- 6 days) - Pulmicort Respules 0.5 mg/mL inhalation suspension: Budesonide 0.5 mg/ml. Each 2 ml Respule contains 1 mg budesonide.
- B/A - Treatment With Pulmicort Respules 1 mg Followed by Treatment With BDA MDI (PT027) 160/180 μg: Subjects randomized to receive a single dose of budesonide by nebulization (Pulmicort Respules) 1mg at Visit 2, and a single dose of budesonide/albuterol by metered-dose inhaler, BDA MDI, (PT027) 160/180 μg at Visit 3.
  Visit 2/Period 1 (Day 1) - Pulmicort Respules 0.5 MG/ML Inhalation Suspension: Budesonide 0.5 mg/ml. Each 2 ml Respule contains 1 mg budesonide.
  Visit 3/Period 2 (Day 8 +/- 6 days) - BDA MDI (PT027) 160/180 μg: Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 80/90 μg per puff. Two puffs to administer 160/180 μg dose.
Period: Period 1 (First Treatment Intervention)
Arm/Group | A/B - Treatment With BDA MDI (PT027) 160/180 μg Followed by Treatment With Pulmicort Respules 1mg | B/A - Treatment With Pulmicort Respules 1 mg Followed by Treatment With BDA MDI (PT027) 160/180 μg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2 (Second Treatment Intervention)
Arm/Group | A/B - Treatment With BDA MDI (PT027) 160/180 μg Followed by Treatment With Pulmicort Respules 1mg | B/A - Treatment With Pulmicort Respules 1 mg Followed by Treatment With BDA MDI (PT027) 160/180 μg
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A/B - Treatment With BDA MDI (PT027) 160/180 μg Followed by Treatment With Pulmicort Respules 1mg | B/A - Treatment With Pulmicort Respules 1 mg Followed by Treatment With BDA MDI (PT027) 160/180 μg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (1.72) | 6.5 (1.64) | 6.2 (1.64)
Age, Customized [Count of Participants; unit: Participants]
  Age group (years): >= 4 to < 6 | 3 | 2 | 5
  Age group (years): >= 6 to <9 | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 4 | 4 | 8
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 118.22 (15.678) | 123.42 (13.939) | 120.82 (14.402)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 26.22 (10.270) | 34.77 (12.430) | 30.49 (11.752)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms per meter squared] | 17.97 (2.641) | 22.07 (3.269) | 20.02 (3.551)

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t
Description: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration
Time Frame: A total of 10 samples were taken per treatment visit at pre-dose and at 10, 20, 40, 60, 120, 240, 360, 480 and 720 minutes after dosing.
Population: Budesonide PK samples were available from 12 children. There were 2 instances, one for each treatment intervention, where the pre-dose budesonide concentration was considered too high (16% and 46% of Cmax), potentially having an impact on the post-dose concentrations. There was also 1 instance in the Pulmicort Respules 1mg treatment intervention where post-dose samples were not collected due to difficulty with the catheter. PK parameters were not calculated in these three instances.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Groups:
- Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects: Individual PK parameters and summary statistics after administration of study treatment A - BDA MDI (PT027) 160/180 μg
- Treatment Intervention B - Pulmicort Respules 1 mg: Individual PK parameters and summary statistics after administration of study treatment B - Pulmicort Respules 1mg
Arm/Group | Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects | Treatment Intervention B - Pulmicort Respules 1 mg
Number analyzed (Participants) | 11 | 10
h*pg/mL | 435 (191) | 1164 (587)

2. Primary Outcome: Cmax
Description: Maximum observed plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects | Treatment Intervention B - Pulmicort Respules 1 mg
Number analyzed (Participants) | 11 | 10
pg/mL | 126 (53.3) | 651 (480)

3. Secondary Outcome: Tmax
Description: Time to reach maximum observed plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects | Treatment Intervention B - Pulmicort Respules 1 mg
Number analyzed (Participants) | 11 | 10
hours | 0.667 [0.333 to 2.00] | 0.167 [0.167 to 0.750]

4. Secondary Outcome: Tlast
Description: Time of last quantifiable plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects | Treatment Intervention B - Pulmicort Respules 1 mg
Number analyzed (Participants) | 11 | 10
hours | 12.0 [8.00 to 12.0] | 12.0 [11.9 to 12.0]

5. Secondary Outcome: Clast
Description: Drug concentration at last observed (quantifiable) concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects | Treatment Intervention B - Pulmicort Respules 1 mg
Number analyzed (Participants) | 11 | 10
pg/mL | 12.5 (5.03) | 18.7 (7.09)

ADVERSE EVENTS:
Time Frame: Approximately one week for each treatment intervention.
Description: Safety population included all subjects who received at least one treatment intervention.
Groups:
- Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects: Safety analysis of subjects receiving Treatment A - BDA MDI (PT027) 160/180 μg
- Treatment Intervention B - Pulmicort Respules 1 mg: Safety analysis of subjects receiving Treatment B - Pulmicort Respules 1mg
Arm/Group | Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects | Treatment Intervention B - Pulmicort Respules 1 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Intervention - BDA MDI (PT027) 160/180 μg - All Subjects (N=12) | Treatment Intervention B - Pulmicort Respules 1 mg (N=12)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
data or results obtained from this study must not be published without prior approval from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT04848662/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT04848662/SAP_001.pdf